CLINICAL TRIAL: NCT00320853
Title: A Pilot Study to Evaluate the Effect of Vitamin D Supplementation on Insulin Secretion and Peripheral Insulin Sensitivity
Brief Title: A Study to Evaluate the Effect of Vitamin D Supplementation on Insulin Sensitivity and Secretion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sitaram Bhartia Institute of Science and Research (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SBISR/2006/02
Record Dates: First submitted 2006-05-01; First posted 2006-05-03 (Estimated); Last update posted 2006-05-03 (Estimated); Status verified 2006-05

CONDITIONS: Diabetes Mellitus, Non-Insulin-Dependent
Keywords: Diabetes; Vitamin D; Insulin sensitivity; Insulin secretion
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Insulin Resistance | interventions — Vitamin D

INTERVENTIONS:
Drug: Vitamin D

SUMMARY:
The purpose of the study is to evaluate the change in insulin sensitivity and secretion indices (early markers for development of diabetes) after 4 weeks of a megadose of Vitamin D. This will also help to calculate sample size for and choose an appropriate index for a larger randomized control trial which may be required subsequently.

DETAILED DESCRIPTION:
Accumulating evidence suggests that serum Vitamin D levels may be inversely related to the prevalence of diabetes, to the concentration of glucose , insulin resistance and metabolic syndrome.The available trials have been conducted using small sample sizes in different subgroups (hemodialyzed patients , healthy volunteers , gestational diabetes and post menopausal women ) document variable results with a positive result in some (hemodialysis and gestational diabetes) and no effect in other settings(healthy volunteers and postmenopausal women).We therefore, planned this trial to study the effect of vitamin D supplementation (240,000 IU) on insulin secretion and peripheral insulin sensitivity.This will also help to calculate sample size for and choose an appropriate index for a larger randomized control trial which may be required subsequently.

Study design and comparison:Single group, open label intervention trial involving assessment of insulin sensitivity and secretion in 30 volunteers before and after 4weeks of a megadose of Vitamin D. The pre and post intervention results will be compared using the paired t test.

ELIGIBILITY:
Inclusion Criteria:

* Male
* ≥30 years of age
* Waist circumference ≥80 cm

Exclusion Criteria:

* Diabetic- Fasting Blood Sugar >126 mg/dl or on anti-diabetic medication
* BP>140/90 or on anti-hypertensive medication
* Receiving Vitamin D or calcium supplementation
* Chronic disease-renal/hepatic/malignancy/gastrointestinal
* On any medication within the last one month which could potentially influence insulin secretion, insulin sensitivity, Vitamin D or Calcium metabolism
* Febrile illness or infective morbidity in the past 10 days

Min Age: 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2006-04; Study Completion 2006-05

PRIMARY OUTCOMES:
OGIS Index, Total Insulin Secretion

SECONDARY OUTCOMES:
HOMA
QUICKI
ISI composite
ISI stumvoll
ISI Gutt
Insulinogenic Index
Lipid profile
CRP
ApoA1
ApoB

CONTACTS AND LOCATIONS:
Overall Officials: Jitendra N Pande, MD, Principal Investigator — Sitaram Bhartia Institute of Science and Research; Jitender Nagpal, MD, Principal Investigator — Sitaram Bhartia Institute of Science and Research; Abhishek Bhartia, ME, Study Director — Sitaram Bhartia Institute of Science and Research; Anupama Singh, MD, Study Chair — Sitaram Bhartia Institute of Science and Research
Locations (1):
- Sitaram Bhartia Institute of Science and Research, New Delhi, National Capital Territory of Delhi, India